CLINICAL TRIAL: NCT00738335
Title: A Phase I Open-Label, Dose-Finding Study to Evaluate the Safety and Efficacy of Concurrent Radiosurgery and Erlotinib Administration in Non-Small Cell Lung Cancer Patients With Brain Metastases
Brief Title: Stereotactic Radiosurgery and Erlotinib in Treating Patients With Non-Small Cell Lung Cancer and Brain Metastases
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000612064; UCSF-072520; CC# 072520; GENENTECH-UCSF-072520
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Lung Cancer; Metastatic Cancer
Keywords: stage IV non-small cell lung cancer; tumors metastatic to brain; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Erlotinib Hydrochloride; Immunoenzyme Techniques; Chromatography, Liquid; Mass Spectrometry; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: erlotinib hydrochloride
Other: immunoenzyme technique
Other: laboratory biomarker analysis
Other: liquid chromatography
Other: mass spectrometry
Other: pharmacological study
Radiation: stereotactic radiosurgery

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Radiation therapy uses high-energy x-rays to kill tumor cells. Stereotactic radiosurgery may be able to deliver x-rays directly to the tumor and cause less damage to normal tissue. Erlotinib may make tumor cells more sensitive to radiation therapy. Giving erlotinib together with stereotactic radiosurgery may kill more tumor cells.

PURPOSE: This phase I clinical trial is studying the side effects of erlotinib when given together with stereotactic radiosurgery and to see how well it works in treating patients with non-small cell lung cancer with brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the acute as well as long-term toxicity (especially grade III neurotoxicity) of concurrent erlotinib hydrochloride and single-fraction radiosurgery in patients with non-small cell lung cancer (NSCLC) and brain metastases.

Secondary

* To determine the freedom from progression in all detected lesions (i.e., radiosurgically treated and untreated) and the rate of response of radiosurgically treated lesions in patients receiving concurrent erlotinib hydrochloride and radiosurgery as compared with historical controls treated with gamma knife radiosurgery alone at UCSF.
* To measure the rate of freedom from any CNS progression in these patients at 1 year post treatment.
* To assess cerebrospinal fluid (CSF) distribution of erlotinib hydrochloride by measuring both erlotinib hydrochloride and its major metabolite, OSI-420, in plasma and CSF at 4 or more days after initial erlotinib hydrochloride administration but before radiosurgery, and again at 4 weeks after stereotactic radiosurgery (optional).
* To perform CSF and serum biomarker analysis for NSCLC using 2-dimensional liquid chromatography or mass spectrometry (2D-LC/MS).
* To determine the incidence of subclinical leptomeningeal disease in patients assigned to gamma-knife treatment and who do not exhibit signs or symptoms or carcinomatous meningitis.

OUTLINE: Patients receive oral erlotinib hydrochloride once daily for at least 7 days. Patients then undergo stereotactic radiosurgery on day 0. Beginning the day after radiosurgery, patients receive erlotinib hydrochloride once daily for 4 weeks in the absence of disease progression or unacceptable toxicity. After completion of study therapy, patients may continue to receive erlotinib hydrochloride at the discretion of their oncologist.

Patients undergo cerebrospinal fluid (CSF) and blood sample collection at baseline (at least 4 days after starting erlotinib hydrochloride and prior to radiosurgery) for pharmacokinetic and biomarker correlative studies. Samples are analyzed for concentrations of erlotinib hydrochloride by 2-dimensional-liquid chromatography/mass spectrometry and antithrombin by enzyme-linked immunosorbent assay.

After completion of study therapy, patients are followed every 3 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer (NSCLC) meeting the following criteria:

  * Fewer than 5 intraparenchymal brain metastases by gadolinium-enhanced MRI meeting the following criteria:

    * Maximum diameter ≤ 4.0 cm

      * If multiple lesions are present and one lesion is > 3.0 cm, the remaining lesions must be ≤ 3.0 cm in maximum diameter
    * No metastases within 3 mm of the optic nerve or optic chiasm such that some portion of the optic nerve or chiasm would receive > 9 Gy from radiosurgery
    * No metastases in the brainstem, midbrain, pons, or medulla
* No prior complete resection of a single brain metastasis or of all known brain metastases

  * Subtotal resection allowed provided residual disease is ≤ 4.0 cm in maximum diameter
* No clinical or radiographic evidence of unstable systemic progression (other than the study lesion[s]) within the past month

  * Patients with brain metastases at initial presentation do not require 1 month of scans documenting stable disease
* Isolated brain metastases with stable systemic disease allowed
* No leptomeningeal metastases by MRI and/or positive cerebrospinal fluid cytology

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Life expectancy ≥ 3 months
* ANC > 1,000/mm³
* Platelet count > 100,000/mm³
* Hemoglobin > 10 g/dL
* PT and PTT normal
* AST < 2 times upper limit of normal (ULN)
* Alkaline phosphatase < 2 times ULN
* Total bilirubin < 2 times ULN
* Lactic dehydrogenase < 2 times ULN
* Serum creatinine < 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 2 weeks after completion of study therapy
* Neurologic function status 0-2
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to erlotinib hydrochloride
* No contraindication to MRI (e.g., cardiac pacemaker)
* No absolute contraindication to lumbar puncture

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior systemic therapy allowed
* No prior cranial radiotherapy

  * Prior radiotherapy to noncranial sites allowed
* More than 1 week since prior intrathecal chemotherapy or prior treatment of leptomeningeal carcinoma
* No concurrent systemic therapy

  * Prior or current erlotinib hydrochloride for treatment of systemic disease allowed provided systemic disease has not progressed while on erlotinib hydrochloride
* No concurrent enzyme-inducing anticonvulsant

  * If patients are on an enzyme-inducing anticonvulsant (e.g., phenytoin, carbamazepine, or phenobarbital), the agent must be converted to a nonenzyme-inducing anticonvulsant before or at the start of erlotinib hydrochloride treatment
* No concurrent CYP3A4 inhibitors or inducers (e.g., Hypericum perforatum [St. John wort] or ketoconazole)
* No other concurrent investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Acute and long-term toxicity (i.e., neurotoxicity, gastrointestinal, cutaneous, and hematologic) as assessed by NCI CTCAE v3.0.

SECONDARY OUTCOMES:
Disease progression
Response rate of radiosurgically treated lesions in patients receiving concurrent erlotinib hydrochloride and radiosurgery on this study vs the response rate of historical controls previously treated with gamma knife radiosurgery alone
CNS progression at 1 year
Distribution of erlotinib hydrochloride in plasma and cerebrospinal fluid (CSF)
CSF and serum biomarkers
Incidence of subclinical leptomeningeal disease

CONTACTS AND LOCATIONS:
Overall Officials: James L. Rubenstein, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States